CLINICAL TRIAL: NCT02366312
Title: A Phase 2, Single-center, Single-arm, Open Label Trial of Vismodegib in Patients With Keratocystic Odontogenic Tumors
Acronym: KCOT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NYU College of Dentistry (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Brian L. Schmidt, Director, Bluestone Center for Clinical Research, NYU College of Dentistry
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-00254; ML28859 (Other: Genentech)
Record Dates: First submitted 2015-02-05; First posted 2015-02-19 (Estimated); Results first posted 2021-02-18 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Keratocystic Odontogenic Tumor
Keywords: Keratocystic odontogenic tumor; KCOT
MeSH Terms: conditions — Odontogenic Cysts | interventions — HhAntag691

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- vismodegib (Experimental): The 150-mg vismodegib drug product is a hard gelatin capsule formulation for oral administration. This study involves one year of treatment with Erivedge (150 mg/day) plus two years of follow-up.
  Interventions: Drug: vismodegib

INTERVENTIONS:
Drug: vismodegib — vismodegib is a synthetic, small molecule inhibitor of the sonic Hh pathway, which is involved in tumorigenesis, thus providing a strong rationale for its use in the treatment of a variety of cancers.
  Other Names: ERIVEDGE®, GDC-0449

SUMMARY:
The purpose of this study is to determine how well a daily dose of 150 mg of Erivedge (vismodegib) reduces Keratocystic odontogenic tumor (KCOT) size, and to evaluate the safety of this dose. Erivedge is FDA-approved for use in adults with a specific type of skin cancer. However, the drug is experimental for patients with KCOT.

DETAILED DESCRIPTION:
This is a single-center, interventional, single-arm, open-label, two-cohort clinical trial. A total of 20 patients will be enrolled (10 with NBCCS-associated KCOT and 10 with sporadic KCOT) over a period of 2 years. This is a 3 year study where each patient will undergo up to 1 year of treatment and up to 2 years of post-treatment follow-up.

All patients will be assessed for safety and efficacy of the study drug GDC-0449 (Vismodegib).

ELIGIBILITY:
Inclusion Criteria:

* Males and females, 18 years of age and above at the time the informed consent form is signed;
* Able to understand and sign the Informed Consent Form and other necessary paperwork prior to initiation of study procedures;
* Able to communicate with the investigator/study site personnel, understand and comply with the study requirements, and willing to return for specified visits at the appointed time;
* Patients who have received prior treatment for their KCOT and with a diagnosis of recurrent (maxillary or mandibular) sporadic KCOT or NBCCS-associated KCOT (single or multiple);
* Diagnosis of KCOT will be done by past pathology report or by biopsy at the study site, if applicable;
* Willingness to consent to biopsy of the lesion, if needed;
* Willingness to delay excision of the target tumor site, unless evidence of disease progression or lack of drug tolerability;
* Willingness to donate blood for genetic testing;
* For female patients of childbearing potential, agreement to use two acceptable methods of birth control, including one barrier method during the study and 7 months after discontinuation of study drug;
* For males with female partners of childbearing potential, agreement to use a male condom (with spermicide) and to advise their female partners to use an acceptable method of birth control during the study and for 2 months after the discontinuation of the study drug;
* Agreement not to donate blood/blood products during the study and for 7 months after the discontinuation of the study drug;
* For males not to donate sperm products or semen during treatment and for 2 months after the discontinuation of the study drug;
* Able and willing to swallow pill;
* No malabsorption syndrome or other condition that would interfere with enteral absorption;
* At least 4 weeks since last chemotherapy, investigational therapy, radiotherapy or major surgical procedure and recovered from the first study drug administration;
* KCOT measures at least 1 cm in one dimension on pretreatment volumetric CT scan;
* No clinically significant abnormalities with clinical laboratory assessments;

Exclusion Criteria:

* Concurrent anti-tumor therapy;
* Completion of the most recent anti-tumor therapy (including Vismodegib) less than 4 weeks prior to the initiation of treatment (first study drug administration);
* Uncontrolled medical illness;
* Pregnancy or lactation; female patients who are planning to become pregnant for the duration of the study and 7 months post-treatment;
* Inability or unwillingness to swallow capsules;
* Any medical or psychological illness or condition preventing adequate consent;
* History of significant atherosclerotic disease, including the following:

  * Coronary artery disease (i.e., myocardial infarction within the past year or unstable angina);
  * Documented carotid atheroma;
* Known HIV infection;
* Current alcohol abuse;
* History of resistance to vismodegib (patients who previous received vismodegib for BCC and had no clinical response will be excluded).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-10-27 (Actual); Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian L Schmidt, DDS, MD, PhD, Principal Investigator — NYU College of Dentistry
Locations (1):
- NYU Bluestone Center For Cllinical Research, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited at the NYU Oral cancer center between mmyy and mmyy. The first participant was enrolled in mmyy and the last subject was enrolled in mmyy.
Pre-assignment Details: Of 3 enrolled subjects, 2 met inclusion criteria and received treatment.
Groups:
- NBCCS-associated KCOT: Nevoid Basal Cell Carcinoma Syndrome (NBCCS)-associated Keratocystic Odontogenic Tumor (KCOT) Group
- Sporadic KCOT: Sporadic Keratocystic Odontogenic Tumor (KCOT) Group
Period: Overall Study
Arm/Group | NBCCS-associated KCOT | Sporadic KCOT
Started | 1 | 1
Completed | 1 | 0 (The subject did not attend the 2-year post-treatment visit (last visit).)
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NBCCS-associated KCOT | Sporadic KCOT | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White - Not Hispanic or Latino | 1 | 0 | 1
  Hispanic or Latino | 0 | 1 | 1
  African American | 0 | 0 | 0
  Asian/Pacific Islander | 0 | 0 | 0
  Other | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 2
Primary KCOT Tumor size at Baseline [Number; unit: centimeter] — Volumetric CT Scan to capture primary KCOT lesion size (greatest dimension) at baseline
  centimeter | 3 | 3.8 | 2

OUTCOME MEASURES:

1. Primary Outcome: KCOT Volume (Greatest Dimension)
Description: To evaluate the efficacy of GDC-0449 in reducing KCOT size (shrinkage) in NBCCS-associated KCOT and sporadic KCOT patients following 6 to 12 months of ingestion of 150 mg/day, up to 1 year of treatment and up to 2 years of post- treatment follow-up.
Time Frame: Baseline, 6 month (in treatment), 1 year (in treatment), 2 Year (post-treatment), 3 Year (post-treatment)
Population: Subjects received ERIVEDGE® (vismodegib) 150 mg capsule orally once daily for 12 months.
Measure: Number; unit: centimeter
Arm/Group | NBCCS-associated KCOT | Sporadic KCOT
Number analyzed (Participants) | 1 | 1
centimeter
  Baseline | 3 | 3.8
  6 month (In treatment) | 0 | 2.6
  1 Year (In treatment) | 2.3 | 2.0
  2 Year (post-treatment) | 2.2 | 1.9
  3 Year (post-treatment) | 2.0 | 0

ADVERSE EVENTS:
Time Frame: Up to three years
Arm/Group | NBCCS-associated KCOT | Sporadic KCOT
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 1/1
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NBCCS-associated KCOT (N=1) | Sporadic KCOT (N=1)
High grade Newuorendocrine Carcinoma of head/neck (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Serious but not related to study drug
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NBCCS-associated KCOT (N=1) | Sporadic KCOT (N=1)
Pain (General disorders) | 0 (0) | 1 (1) — Right jaw pain / non serious / possibly related
Earache (Ear and labyrinth disorders) | 0 (0) | 1 (1) — Non-serious / unlikely related
Sore Throat (General disorders) | 0 (0) | 1 (1) — non-serious / unlikely related
Cramping (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Right hand cramping / non-serious / possibly related to study drug
spasm (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Left Quadricep Spasm / non-serious / probably related to study drug
Allergic reaction (General disorders) | 1 (1) | 0 (0) — right face / non-serious / not related
Spasm (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Both legs / non-serious / probably related
cramp (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — finger cramping / non-serious / probably related
Hair loss (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — non-serious / possibly related
Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) — epigastric pain / non-serious / unlikely related
Facial numbness (Nervous system disorders) | 1 (1) | 0 (0) — Right side / non-serious / probably related
Leg Cramp (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — worsening of leg cramps / non-serious / probably related
Chest Discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) — non-serious / not related / possible related
Cold symptoms (General disorders) | 1 (2) | 0 (0) — non-serious / not related
GI upset (Gastrointestinal disorders) | 1 (2) | 0 (0) — Non serious / Not related / possibly related
Upper Respiratory Infection (Reproductive system and breast disorders) | 1 (1) | 0 (0) — non-serious / unlikely related
Loss of taste (General disorders) | 0 (0) | 1 (1) — non-serious, possibly related
Toes cramping (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — non-serious, possible related
Loose stool (Gastrointestinal disorders) | 1 (2) | 0 (0) — non-serious, possible related
lower extremity pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — both sides, non-serious, possibly related
Right facial pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — non serious, possibly related
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Left sided muscle ache (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — non-serious, not related
Sacral injury (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — non-serious , not related
Nasopharyn lesion (Infections and infestations) | 0 (0) | 1 (1) — non serious, possibly related
bilateral lower extremities swelling (Endocrine disorders) | 0 (0) | 1 (1) — non-serious , unlikely related

LIMITATIONS AND CAVEATS:
Enrollment for the study closed early by the sponsor due to low enrollment number. Only two subjects were enrolled and received the study treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-10-14): https://cdn.clinicaltrials.gov/large-docs/12/NCT02366312/Prot_SAP_000.pdf
  • Informed Consent Form (2016-10-20): https://cdn.clinicaltrials.gov/large-docs/12/NCT02366312/ICF_001.pdf